CLINICAL TRIAL: NCT05054868
Title: Effect of Ketorolac Administration on Post-operative Narcotic Utilization and Union Rates in Great Toe Arthrodesis
Brief Title: Ketorolac vs Oxycodone for Great Toe Arthrodesis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001123
Record Dates: First submitted 2021-07-23; First posted 2021-09-23 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Arthrodesis
Keywords: big toe arthrodesis; big toe; joint fusion
MeSH Terms: conditions — Ankylosis | interventions — Oxycodone; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Control group) - Oxycodone only (Active Comparator): Subjects randomized to this group will receive oxycodone for postop pain management (standard of care).
  Interventions: Drug: Oxycodone
- Group 2 (Treatment group) - Oxycodone and Ketorolac (Experimental): Subjects randomized to this group will receive oxycodone and ketorolac for postop pain management.
  Interventions: Drug: Oxycodone; Drug: Ketorolac

INTERVENTIONS:
Drug: Oxycodone — Subjects randomized to the control group will receive oxycodone for postop pain management (standard of care).
Drug: Ketorolac — Subjects randomized to the treatment group will receive oxycodone and ketorolac for postop pain management.
  Arms: Group 2 (Treatment group) - Oxycodone and Ketorolac

SUMMARY:
This study reviews if taking ketorolac, after a joint fusion procedure, can decrease the need for taking oxycodone (standard of care) for pain relief. The study also investigates if ketorolac affects bone healing after surgery.

DETAILED DESCRIPTION:
This study reviews if taking ketorolac, after a joint fusion procedure, can decrease the need for taking oxycodone (standard of care) for pain relief. The study also investigates if ketorolac affects bone healing after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years.
* Women of childbearing potential must have a negative serum or urine pregnancy test results within 24 hours before the first dose of ketorolac.
* Primary elective great toe MTP arthrodesis (CPT 28750). Other forefoot procedures often performed in conjunction with toe fusion will be included (CPT codes 28308, 28285, 28270).

Exclusion Criteria:

* Chronic pain syndrome, CRPS or fibromyalgia
* Revision procedures
* Use of allograft bone at the fusion site
* Tobacco use
* Diabetes
* Narcotic abuse or IV drug abuse
* Any CPT codes involving the midfoot, hindfoot, and/or ankle
* Unable to take NSAIDs secondary to medical comorbidities such as kidney disease (impaired renal function with CrCl ≤ 50 ml/min) or gastric ulcers
* Weight < 50 kg
* Does not speak or read English
* If pregnant or planning to become pregnant or breastfeeding
* Non-independent dweller (prisoner)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-04-14 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain scores - collected at baseline (standard of care) and for the study using a study survey on days 3, 7, and 14 after surgery. | From baseline to 14 days after the surgery
  To study if postop ketorolac provides effective pain relief and helps reduce the need to take oxycodone. Participants will complete a short survey on Days 3, 7, and 14 after surgery. Participants will be asked to provide VAS pain scores, on a scale of 1-10, for the past 24 hours on Days 3, 7, and 14 after surgery.
Quantitative pain management - measured using a study survey. | 14 days after the surgery
  To study if postop ketorolac provides effective pain relief and helps reduce the need to take oxycodone. Participants will complete a short survey on Days 3, 7, and 14 after surgery. The survey will ask the following set of questions-
  * number of pills (oxycodone and/or ketorolac) consumed
  * if the pain medicine(s) needed to be refilled
  * discontinuation date & reason
  * side effects, if any
  * the effectiveness of the pain medicine(s)
  * preference for ketorolac or oxycodone, if applicable

OTHER OUTCOMES:
Bone fusion - doctor will review the 3 month postop x-ray to see if the bones have fused at the site of surgery | Approximately 90 days after surgery (or until 3-month post-op visit is completed)
  To study if postop ketorolac affects bone fusion. This will be assessed by comparing the routine x-rays collected at the baseline visit to the routine x-rays taken at the 3-month postop visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Amy Loveland, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No